CLINICAL TRIAL: NCT05017441
Title: TOcilizumab and Covid-19 : Risk of Severe INfection
Acronym: TOCSIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: TOCSIN
Record Dates: First submitted 2021-08-19; First posted 2021-08-23 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SARS-CoV2 is responsible for a pandemic that has been evolving for approximately 18 months. The virus' capacity for dissemination and its virulence are responsible for significant morbidity and mortality. The initial lack of knowledge of the pathogen and of the pathophysiology underlying the potential severity of the disease, particularly in the respiratory tract, led to numerous therapeutic attempts in this emergency context, centered on the control of an obviously exaggerated inflammatory response. A large number of studies remained of insufficient quality to lead to relevant and applicable conclusions. Secondly, the benefit of corticosteroid therapy has been demonstrated in two trials. Although Dexamethasone remains the only corticosteroid to improve survival, these results have reinforced the hypothesis of the interest of treatments reducing the inflammatory response, particularly cytokine. The widespread use, in the absence of scientific data, of interleukin-6 receptor inhibitors (Sarilumab and Tocilizumab) has been structured around studies whose results remain uncertain to this day because of the heterogeneity of the population treated and the results observed. A possible survival benefit seems to emerge for resuscitation patients who have not yet required invasive ventilation, the other situations being probably associated with the absence of effect or even the potential danger of this treatment. Tocilizumab is notably associated in the literature with the risk of secondary infections and mucosal healing abnormalities, favoring bleeding complications and digestive perforations. The objective of this study is to evaluate the risk of digestive complications (hemorrhage, perforation, diverticulitis) and infectious complications related to the use of Tocilizumab according to the severity of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* French-speaking patient
* Patient with COVID-19 documented by PCR test or chest CT scan

Exclusion Criteria:

* No confirmation of suspected COVID-19
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his/her data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with COVID-19 documented by PCR test or chest CT scan, treated in hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of infectious episodes during the hospitalization period | Day 90
  This outcome corresponds to occurrence of an infectious episode during hospitalization in a ward and/or intensive care unit.

SECONDARY OUTCOMES:
Digestive complication rate | Day 90
  This outcome corresponds to the number of patients who had digestive complications.
Rate of hematological complications | Day 90
  This outcome corresponds to the number of patients who had hematological complications.
Death rates | Day 90
  This outcome corresponds to the number of patients who died at D90.
Death rates | Day 28
  This outcome corresponds to the number of patients who died At D28.

CONTACTS AND LOCATIONS:
Overall Officials: François PHILIPPART, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Birgand G, Peiffer-Smadja N, Fournier S, Kerneis S, Lescure FX, Lucet JC. Assessment of Air Contamination by SARS-CoV-2 in Hospital Settings. JAMA Netw Open. 2020 Dec 1;3(12):e2033232. doi: 10.1001/jamanetworkopen.2020.33232. PMID 33355679
- [Background] Ong SWX, Tan YK, Chia PY, Lee TH, Ng OT, Wong MSY, Marimuthu K. Air, Surface Environmental, and Personal Protective Equipment Contamination by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) From a Symptomatic Patient. JAMA. 2020 Apr 28;323(16):1610-1612. doi: 10.1001/jama.2020.3227. PMID 32129805
- [Background] Leung NHL. Transmissibility and transmission of respiratory viruses. Nat Rev Microbiol. 2021 Aug;19(8):528-545. doi: 10.1038/s41579-021-00535-6. Epub 2021 Mar 22. PMID 33753932
- [Background] KENDALL EJ, BYNOE ML, TYRRELL DA. Virus isolations from common colds occurring in a residential school. Br Med J. 1962 Jul 14;2(5297):82-6. doi: 10.1136/bmj.2.5297.82. No abstract available. PMID 14455113
- [Background] Yin Y, Wunderink RG. MERS, SARS and other coronaviruses as causes of pneumonia. Respirology. 2018 Feb;23(2):130-137. doi: 10.1111/resp.13196. Epub 2017 Oct 20. PMID 29052924
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Derived] Lefevre C, Funck-Brentano T, Cachanado M, Plocque A, Youinou M, Fels A, Pene F, Savale L, Montani D, Voisin O, Bintein F, Wildenberg L, Philippe A, Legriel S, Roche N, Burgel PR, Tran M, Noel N, Baillard C, Duranteau J, Chatellier G, Philippart F. Benefit and risk associated with interleukin-6 receptor inhibitor administration during severe COVID-19: a retrospective multicentric study. Sci Rep. 2026 Jan 22. doi: 10.1038/s41598-026-36864-w. Online ahead of print. PMID 41571778
- [Derived] Sandhu G, Piraino ST, Piticaru J. Secondary Infection Risk in Patients With Severe COVID-19 Pneumonia Treated With Tocilizumab. Am J Ther. 2022 May-Jun 01;29(3):e275-e278. doi: 10.1097/MJT.0000000000001487. Epub 2022 Mar 4. PMID 35249968